CLINICAL TRIAL: NCT07262242
Title: Comparing Effect of Opioid-sparing Versus Conventional Anesthesia on Quality of Recovery After Emergency Laparotomy: a Randomized Controlled Trial
Brief Title: Effect of Opioid-sparing Anesthesia on Quality of Recovery After Emergency Laparotomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Hasanin, Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MD-5-2025
Record Dates: First submitted 2025-11-17; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Emergency Abdominal Surgery; Opioid Sparing Anaesthesia
MeSH Terms: interventions — Lidocaine; Pharmaceutical Preparations; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lidocaine group (Active Comparator): lidocaine bolus at induction followed by infusion until the end of procedure
  Interventions: Drug: Lidocaine (drug)
- Fentanyl group (Active Comparator): fentanyl bolus at induction followed by saline infusion until the end of procedure
  Interventions: Drug: Fentanyl (IV)

INTERVENTIONS:
Drug: Lidocaine (drug) — induction bolus of 0.15 mL/kg of 10mg/ml lidocaine, followed by 0.15 mL/kg/h infusion (10 mg/mL lidocaine) until end of procedure
  Arms: lidocaine group
Drug: Fentanyl (IV) — induction bolus of 0.15 mL/kg of 10mg/ml fentanyl, followed by 0.15 mL/kg/h infusion (saline) until end of procedure
  Arms: Fentanyl group

SUMMARY:
Opioids are widely used during anesthesia for pain control, but they cause many side effects-such as nausea, constipation, respiratory depression, dependence, and delayed recovery. They can also worsen low blood pressure in patients with unstable circulation. Because of these risks, multimodal analgesia is recommended to reduce opioid use.

Research on other non-opioid options is limited. Systemic lidocaine offers anti-inflammatory and opioid-sparing benefits and improves recovery in elective colorectal surgery, but its role in emergency laparotomy is still unclear and requires further study.

DETAILED DESCRIPTION:
Upon arrival to the operating room, routine monitors will be applied; intravenous line will be secured, and 8 mg dexamethasone will be slowly administrated. Baseline preoperative blood pressure will be recorded as the average of three readings with difference less than 5 mmHg.

Preoperative fluid management Fluid responsiveness will be defined as a 10% increase in stroke volume after passive leg raising maneuver. Fluid responder will be given 500-mL bolus of lactated ringer. Passive leg raising will be repeated until wither the patient is non-responder or 1500 mL were infused.

induction of anesthesia: 2 mg/kg propofol and 1 mg/kg succinyl choline. Anesthesia will be maintained by isoflurane in air/oxygen admixture (with target end tidal isoflurane 1-1.2%). Atracurium will be administered after patient recovery from succinylcholine at a dose of 0.5 mg/Kg and then regularly according to local protocols.

A 10-12 mL/kg/hr of lactated ringer will be infused during the procedure. Heart rate and blood pressure will be monitored at 2 min intervals. The average of every 5 successive readings would be recorded every 10 min. If patients developed hypotension (mean arterial pressure (MAP) ≤ 70% of the baseline reading and/or <65 mmHg), a fluid bolus of 4 mL/kg will be given and the change in the pulse pressure will be noted. If the pulse pressure increases by >10 %, the fluid bolus will be given until the increase in pulse pressure is <10%. If hypotension persists despite the adequate volume replacement a 5-mcg bolus of norepinephrine will be given. The bolus will be repeated if MAP was not restored within 2 min. Infusion of norepinephrine can be given if MAP persisted <65 mmHg despite 5 boluses of norepinephrine.

If bradycardia occurred (defined as heart rate less than 55 bpm), it will be managed by IV atropine bolus (0.5 mg).

Intraoperative tachycardia and/or hypertension (defined as 20% increase from the baseline value) will be managed by fentanyl bolus of 0.5 mcg/kg, in absence of other causes.

At the end of the procedure, all patients will receive 1 gm of paracetamol intravenously and local infiltration of the wound with 40 mL of 0.125% bupivacaine. Patients who are not indicated for extubation at the end of the surgery will be excluded from the study.

Postoperative management All patients will receive 1 gm/ 6h of paracetamol. Static (at rest) and dynamic (during cough) numerical rating scale (NRS) will be assessed at 0.5, 2, 6, 10, 16, 24 hr postoperatively. If the NRS>3, a 2 mg morphine bolus will be given to be repeated after 30 min if pain persists.

4 mg of ondansetron will be given if patients developed nausea or vomiting.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (21-65 years), ASA I-III undergoing emergency laparotomy with midline incision

Exclusion Criteria:

* Severe cardiac morbidities (impaired contractility with ejection fraction < 45%, heart block, arrhythmias, tight valvular lesions)
* Patients on vasopressor infusion, patients with high shock index (heart rate / systolic blood pressure >1)
* Body mass index <18 or > 35 Kg/m2,
* Pregnant or lactating women,
* Allergy of any of the study drugs
* Severe liver cell failure and renal impairment by history and/or abnormal liver and kidney function tests.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Quality of recovery using QoR-15 | 24 hours after surgery
  The QoR-15 scale is a global measure of postoperative recovery, with a score ranging from 0 (extremely poor QoR) to 150 (excellent QoR)

SECONDARY OUTCOMES:
intraoperative fentanyl consumption | from time of induction of anesthesia until end of procedure
  mcg/kg
mean arterial pressure | at baseline preoperatively, every 10 minutes (averaging of each 5 readings) from induction of anesthesia until end of procedure, and 2, 6, 10, 16, 24 hours postoperatively.
  mmHg
heart rate | at baseline preoperatively, every 10 minutes (averaging of each 5 readings) from induction of anesthesia until end of procedure, and 2, 6, 10, 16, 24 hours postoperatively.
  bpm
postoperative opioid consumption | from extubation until 24 hours postoperatively
  nalbuphine in mg
numeric rating scale | 30 minutes, 2-, 6-, 10-, 16-, 24 hours postoperatively
  rate pain on a scale of 0-10, 0: no pain, 10: worst pain
serum lactate | 30 minutes postoperative
respiratory rate | 30 minutes postoperative
Oxygen saturation/ fraction of inspired oxygen (SF ratio) | 30 minutes postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alainy Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
data related to this research are available from the PI upon reasonable request